CLINICAL TRIAL: NCT04709887
Title: Appropriate Strategy of Surgical Treatment in Ischemic Diabetic Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Hailin Xu, Associate Professor, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mTTTDFU01
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Foot; Ischemic Diabetic Foot Ulcer; Popliteal Artery Stenosis
Keywords: Ischemic Diabetic Foot Ulcer; Surgical Strategy; Cohort study
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Rate of popliteal artery stenosis < 50%, W. (Other): If the rate of popliteal artery stenosis of patients < 50%, the patients only receive the wound treatment.
  Interventions: Procedure: Wound treatment
- Rate of popliteal artery stenosis < 50%, WT. (Other): If the rate of popliteal artery stenosis of patients < 50%, the patients receive the wound treatment and tibial transverse transport surgery.
  Interventions: Procedure: Wound treatment; Procedure: Tibial transverse transport surgery
- Rate of popliteal artery stenosis ≥ 50%, WV. (Other): If the rate of popliteal artery stenosis of patients ≥ 50%, the patients receive the wound treatment and vascular intervention surgery.
  Interventions: Procedure: Wound treatment; Procedure: Vascular intervention surgery
- Rate of popliteal artery stenosis ≥ 50%, WT. (Other): If the rate of popliteal artery stenosis of patients ≥ 50%, the patients receive the wound treatment and tibial transverse transport surgery.
  Interventions: Procedure: Wound treatment; Procedure: Tibial transverse transport surgery
- Rate of popliteal artery stenosis ≥ 50%, WVT. (Other): If the rate of popliteal artery stenosis of patients ≥ 50%, the patients receive the wound treatment, vascular intervention and tibial transverse transport surgery.
  Interventions: Procedure: Wound treatment; Procedure: Vascular intervention surgery; Procedure: Tibial transverse transport surgery

INTERVENTIONS:
Procedure: Wound treatment — According to the guidelines and recommendations of the International Diabetic Foot Working Group, ulcer surface debridement, negative pressure suction drainage, and routine dressing were performed until the wound healed or the end of the trial.
Procedure: Vascular intervention surgery — Segmented distal angiography under the guidance of digital subtraction angiography (DSA) were perform after local anesthesia. The superficial artery is expanded by a 3-4 mm balloon.
  Arms: Rate of popliteal artery stenosis ≥ 50%, WV.; Rate of popliteal artery stenosis ≥ 50%, WVT.
Procedure: Tibial transverse transport surgery — In the anteromedial area of the proximal tibia of the affected limb, the external fixation frame was compared with the area along the midline of the medial longitudinal axis of the proximal tibia. Subsequently, two 3.0 Steinmann pins were inserted through the single layer of cortical bone. The skin was cut along the long axis with the 3.0 Steinmann pin as the centre, and the subcutaneous tissue was separate bluntly to expose the periosteum. The Steinmann pins were used as the centre point for the drilling on four sides with a 2.0 drill bit and use of a rapid osteotomy device; the length of each side was 2.5 cm. Subperiosteal osteotomy was performed with a 5-mm narrow bone knife at an angle of 15°-30° to the bone surface. The surgeons should pay attention to protect the blood supply of the periosteum during this procedure. The external fixators were fixed with 4.0 Steinmann pins at the distal and proximal ends. The subcutaneous tissue and skin were sutured.
  Arms: Rate of popliteal artery stenosis < 50%, WT.; Rate of popliteal artery stenosis ≥ 50%, WT.; Rate of popliteal artery stenosis ≥ 50%, WVT.

SUMMARY:
This cohort study aims to evaluate the outcomes of appropriate surgical treatment strategies in diabetic foot ulcers with different rate of popliteal artery stenosis(<50% or ≥50%). In this study, patients with Texas university grade 2-4(stage C-D) ischemic diabetic foot ulcers will be included. Data of patients who underwent surgical treatment in the past will be retrospectively collected. The patients with follow-up time less than 12 months will continue to follow up. Also the postoperative patients will be prospectively collected. Effects of different surgical strategies, including wound healing therapy, interventional therapy and tibial transverse bone transport therapy will be measured by several indexes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic foot, according to "Chinese Guidelines for Diagnosis and Treatment of Diabetic Foot (2017)".
* Texas university grade 2-4(stage C-D) ischemic diabetic foot ulcers.
* Have clear consciousness, not suffer from mental illness, can cooperate in research and treatment.
* Patients who are informed, participate in the research voluntarily, and have signed the informed consent.
* Have complete clinical data.

Exclusion Criteria:

* Patients with severe systemic infection, who need to be amputated immediately to save lives.
* Patients with mental illness, who cannot cooperate to complete the adjustment and nursing of the external fixator.
* Patients with severe cardiovascular and cerebrovascular diseases (such as severe cardiac insufficiency, severe sequelae of cerebrovascular disease), or with acute infectious diseases.
* Have used or using glucocorticoids systemically within 3 months before admission.
* Have participated in other medical clinical trials within 3 months before admission.
* Patients with severe liver or kidney function abnormalities
* Pregnant or lactating women.
* Patients who lost follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Healing rate of wound surface | 12 months after surgical operation

SECONDARY OUTCOMES:
Ankle-brachial index | 3 months after surgical operation
Ankle-brachial index | 12 months after surgical operation
Recurrence rate of foot ulcer | 12 months after surgical operation

CONTACTS AND LOCATIONS:
Overall Officials: Hailin Xu, MD, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China